CLINICAL TRIAL: NCT05359796
Title: Clinical Characteristics of People With Long-term Type 1 Diabetes: a Cohort Study
Brief Title: Clinical Characteristics of People With Long-term Type 1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Xia Li, Professor, Department of Endocrinology, Institute of of Metabolism and Endocrinology, Nationa Clinical Research Center for Metabolic Diseases, Second Xiangya Hospital of Central South University, Second Xiangya Hospital of Central South University
Other Study IDs: long-term T1D 2022
Record Dates: First submitted 2022-04-24; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Genetic Variation; Functional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, peripheral blood mononuclear cells, urine, feces, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- long-term T1D: Subjects who has the T1D duration ≥10 years, with or without diabetic complications.
  Interventions: Biological: Chronic hyperglycemia; Biological: Residual islet function; Genetic: Genetic variation; Dietary Supplement: Dietary constitutes; Genetic: Microbiome composition and function; Biological: Metabolome composition; Biological: Composition of peripheral blood immune cells

INTERVENTIONS:
Biological: Chronic hyperglycemia — For each follow-up, the glycated albumin(GA) reflecting glycemic control of the past 2-3 weeks, the glycated hemoglobin(HbA1c) reflecting glycemic control of the past 2-3 months, and the advanced glycation end products(AGEs) will be measured.
Biological: Residual islet function — For each follow-up, fasting and stimulated C-peptide levels will be measured.
Genetic: Genetic variation — Genetic variations of interest will be detected with the blood sample collected at baseline.
Dietary Supplement: Dietary constitutes — For each follow-up, the dietary constitutes for the past 3 days will be recorded.
Genetic: Microbiome composition and function — For each follow-up, the fecal and oral samples will be collected for measurement.
Biological: Metabolome composition — For each follow-up, the serum and urine samples will be collected for measurement.
Biological: Composition of peripheral blood immune cells — For each follow-up, the peripheral blood mononuclear cells will be collected for measurement.

SUMMARY:
Type 1 diabetes (T1D) is characterized by absolute insulin deficiency. Although the discovery and application of exogenous insulin has prolonged the lifespan of T1D patients, the chronic diabetic complications caused by long-term poor glycemic control will still reduce patients' quality of life and the overall life expectancy. According to the studies focused on long-term T1D, part of the patients with long disease duration showed resistance to microvascular complications, and several protective factors have been identified. The prevalence of T1D in China is extremely low compared to that in the western world, and little is known about the characteristics of patients with long-term T1D in China. Therefore, this study is designed to collect variable clinical and laboratory features of patients with long-term T1D, explore the risk and protective factors for the development of microvascular complications, and provide reference for the prediction and prevention of these complications.

DETAILED DESCRIPTION:
This is a single-center, prospective, observational study. The investigators propose to enroll 400 patients with type 1 diabetes (T1D) ≥10 years. The patients will be followed up annually for 3 years.

In order to ensure high quality data, two staff are responsible for the input of original data into the database to check and confirm the accuracy. When the data entered by two people is inconsistent, the auxiliary staff decides which data to use.

Missing data will be filled in with the multiple imputation method. The regression analysis will be used to explore the risk and protective factors for the development and progression of microvascular complications.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with type 1 diabetes(T1D) according to the 1999 World Health Organization report
* Insulin dependence from disease onset
* with T1D duration of ≥10 years
* able to understand the procedures and methods of this study, voluntarily participate in the study, and agree to sign the informed consent form

Exclusion Criteria:

* patients with type 2 diabetes, gestational diabetes, or specific types of diabetes
* patients with mental disability or have any other condition or disease that may hamper compliance with the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: subjects are enrolled from hospital, primary care clinic, or community of the whole country
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
the development or progression of diabetic nephropathy | from May 2022 to December 2025
  measured by urine microalbumin/creatinine
the development or progression of diabetic retinopathy | from May 2022 to December 2025
  diagnosed by an ophthalmologist based on fundus photography

SECONDARY OUTCOMES:
the changes of memory function | from May 2022 to December 2025
  measured by the Auditory Verbal Learning Test (AVLT)
the changes of executive function | from May 2022 to December 2025
  measured by the Shape Trail Test (STT)
the changes of language function | from May 2022 to December 2025
  measured by the Boston Naming Test (BNT)
the changes on magnetic resonance imaging(MRI) | from May 2022 to December 2025
  the MRI reflects the changes of cerebral structure and functional connectivity
the changes of bone mineral density(BMD) | from May 2022 to December 2025
  measured by dual x-ray absorbtiometry(DXA), indicating bone density
the changes of brachial-ankle pulse wave velocity(baPWV) | from May 2022 to December 2025
  measured by ultrasound, indicating large artery stiffness
the changes of carotid intima-media thickness(IMT) | from May 2022 to December 2025
  measured by ultrasound, indicating the form of carotid atherosclerotic plaque

CONTACTS AND LOCATIONS:
Overall Officials: Xia Li, MD/PHD, Principal Investigator — Central South University
Locations (1):
- Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No